CLINICAL TRIAL: NCT07185776
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of HRS-5632 Injection in Adult Patients at High Risk of Cardiovascular Events With Elevated Lipoprotein(a)
Brief Title: A Study of HRS-5632 in Adult Participants With Elevated Lipoprotein(a) at High Risk for Cardiovascular Events
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5632-201
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Lipoprotein Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HRS-5632 Dose 1 Group (Experimental)
  Interventions: Drug: HRS-5632 Injection
- HRS-5632 Dose 2 Group (Experimental)
  Interventions: Drug: HRS-5632 Injection
- HRS-5632 Dose 3 Group (Experimental)
  Interventions: Drug: HRS-5632 Injection
- HRS-5632 Dose 4 Group (Experimental)
  Interventions: Drug: HRS-5632 Injection
- HRS-5632 Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-5632 Injection Placebo

INTERVENTIONS:
Drug: HRS-5632 Injection — HRS-5632 injection.
  Arms: HRS-5632 Dose 1 Group; HRS-5632 Dose 2 Group; HRS-5632 Dose 3 Group; HRS-5632 Dose 4 Group
Drug: HRS-5632 Injection Placebo — HRS-5632 injection placebo.
  Arms: HRS-5632 Placebo Group

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of HRS-5632 in adult participants with elevated Lipoprotein(a) (Lp(a)) at high risk for cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the specific procedures of the trial, voluntarily participating in this trial, and providing written informed consent;
2. Being at least 18 years of age on the day of signing the informed consent form;
3. Body Mass Index (BMI) within the range of 18.5 to 40 kg/m² (inclusive of boundary values);
4. Participants must be at high risk of cardiovascular events, defined as individuals diagnosed with Atherosclerotic Cardiovascular Disease (ASCVD) and those at moderate risk or high risk for ASCVD；
5. Based on clinical practice, participants receiving the following medications must be receiving a stable regimen prior to screening or randomization and expected to remain on a stable regimen at the end of the treatment follow-up period:

   1. Lipid-lowering drugs (statins, cholesterol absorption inhibitors, prescription-dose niacin, fibrates, fish oil or other omega-3 fatty acid-containing products, including over-the-counter [OTC] preparations) must be receiving a stable regimen for ≥ 8 weeks prior to randomization; PCSK9 monoclonal antibodies must be receiving a stable regimen for ≥ 12 weeks prior to screening;
   2. Testosterone, estrogen, anti-estrogen/anti-androgen, progestin, selective estrogen receptor modulator, or growth hormone must be receiving a stable regimen for ≥ 4 weeks prior to screening;
6. Participants (including their partners) are willing to voluntarily use highly effective contraceptive measures from the time of signing the informed consent form until 1 year after the last administration of the study drug; female participants must have a negative blood pregnancy test and must not be breastfeeding;
7. Willing and able to comply with all the provisions of the protocol, including demonstrating the ability to adhere to study procedures prior to random assignment.

Exclusion Criteria:

1. Any of the following events occurring within 3 months prior to screening or between screening and randomization, or other events considered by the investigator to indicate clinical instability: major cardiac or non-cardiac surgery; coronary, carotid, or peripheral arterial revascularization; stroke or transient ischemic attack, myocardial infarction or unstable angina, acute limb ischemia, and uncontrolled arrhythmias requiring treatment;
2. Cardiac, cerebrovascular, or peripheral arterial surgery or coronary revascularization planned or anticipated during the trial after randomization;
3. A history of hemorrhagic stroke or other major bleeding (e.g., hemophilia, von Willebrand disease, coagulation factor deficiency), or a hemorrhagic stroke or other major bleeding event (fatal; major organ bleeding; resulting in a rapid, short-term decrease in hemoglobin or blood transfusion) occurring between the screening visit and the randomization visit;
4. Patients with an indication for anticoagulation at screening but not receiving anticoagulation therapy, such as patients with atrial fibrillation or flutter or those undergoing aortic valve replacement;
5. History of any organ system malignancy within 5 years prior to screening (excluding cured basal cell or squamous cell skin cancer, non-invasive stage 0 cervical cancer, non-invasive stage 0 prostate cancer, or ductal carcinoma in situ of the breast), or a history of any organ system malignancy diagnosed between the screening visit and the randomization visit, regardless of whether there is evidence of local recurrence or metastasis;
6. A history of a disease that significantly affects lipid levels, such as nephrotic syndrome, severe liver disease, or Cushing's syndrome;
7. Uncontrolled type 1 or type 2 diabetes (including diabetic ketoacidosis or hyperglycemic hyperosmolar state) within 6 months prior to screening, or HbA1c > 8.0% at screening (secondary confirmation is permitted);
8. History of acute kidney injury within 12 months prior to screening;
9. Uncontrolled hyperthyroidism or hypothyroidism at screening or before randomization;
10. Active infection requiring systemic antiviral or antibacterial medication before randomization;
11. New York Heart Association (NYHA) class III-IV heart function or a most recently measured left ventricular ejection fraction (LVEF) <30% at screening or before randomization;
12. At screening or before randomization, patients, as determined by the investigator, have a major medical condition that is currently unstable and not adequately controlled, such as hematologic disease, renal disease, metabolic or endocrine dysfunction, gastrointestinal disease, chronic disease or infection, unstable mental health disorder, or are recovering from major surgery;
13. Long-term continuous or repeated use of systemic corticosteroids within 3 months prior to screening (excluding local use, such as intra-articular, nasal, inhaled, topical, etc.; long-term continuous means ≥ 7 days; repeated means cumulative use ≥ 3 times);
14. Lipoprotein apheresis within 3 months prior to screening, or plans to undergo such treatment during the study;
15. Patients who are allergic to the active ingredient or any excipients of HRS-5632;
16. Uncontrolled hypertension (sitting systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) before randomization;
17. eGFR < 30 ml/min/1.73 m² (calculated using the CKD-EPI 2009 formula) at screening or before randomization, or current dialysis;
18. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma-glutamyltransferase (GGT) more than 3 times the upper limit of normal (ULN), or total bilirubin more than 1.5 times the ULN at screening or before randomization;
19. Fasting triglycerides ≥ 5.6 mmol/L before randomization;
20. HIV infection (HIV-Ab positive), hepatitis C virus infection (HCV-RNA positive), Treponema pallidum infection (Treponema pallidum antibody positive), or hepatitis B virus infection (HBsAg or HBV-DNA positive) at screening or before randomization;
21. Creatine kinase (CK) levels more than 3 times the ULN before randomization;
22. Thyroid-stimulating hormone (TSH) levels below the lower limit of normal (LLN) or more than 1.5 times the ULN before randomization;
23. Significant abnormalities in laboratory test indicators at screening or before randomization, deemed unsuitable for participation in this study by the investigator;
24. Recent history (within the past year) of drug or alcohol abuse or dependence;
25. Pregnant or breastfeeding women;
26. Participants who have participated in any drug or medical device clinical trial within 3 months prior to screening (participation in a clinical trial is defined as the participant receiving treatment with the investigational drug/device), or who have been exposed to the investigational drug for less than 5 half-lives before screening, whichever is longer;
27. Participants who, as determined by the investigator, are noncompliant or have any other factors that make them unsuitable for participation in the trial, including but not limited to participation that would place the participant at unacceptable risk or could interfere with study evaluations, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The percent change from the baseline in Lipoprotein (a) (Lp(a)). | From baseline to Day 360.

SECONDARY OUTCOMES:
The percentage of all reported adverse events (AEs). | From Day 1 to Day 540.
The percentage of all reported serious adverse events (SAEs). | From Day 1 to Day 540.
The percentage of treatment-related adverse events. | From Day 1 to Day 540.
The percentage of treatment-related serious adverse events. | From Day 1 to Day 540.
The percentage of participants achieving Lipoprotein(a) (Lp(a)) < 125 Nanomole/Liter (nmol/L). | Day 540.
The percentage of participants achieving Lipoprotein(a) (Lp(a)) < 75 Nanomole/Liter (nmol/L). | Day 540.
The plasma concentration of HRS-5632. | From Day 1 to Day 540.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of AFMU, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided